CLINICAL TRIAL: NCT03953066
Title: The Comparison of Serum and Colostral Melatonin, and IL-6 Levels Between Women With Vaginal Delivery, Emergency Cesarean Section and Elective Cesarean Section
Brief Title: Colostral Milk and Blood IL-6 Levels in Types of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, canan soyer çalışkan, MD, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SamsunERH-1
Record Dates: First submitted 2019-04-11; First posted 2019-05-16 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Indications for Care in Pregnancy; Labor; and Delivery
Keywords: melatonin,colostral milk,IL-6, delivery, cesarean section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- women with vaginal delivery (Active Comparator): 30 women with spontaneous vaginal delivery will be included in group 1 serum IL-6 levels before and after delivery and colostral milk melatonin levels will be measured
  Interventions: Other: The calculation of blood IL-6 and coloctral milk melatonin
- women with emergency cesarean section (Active Comparator): 30 women with emergency cesarean section will be included in group 2 serum IL-6 levels before and after delivery and colostral milk melatonin levels will be measured
  Interventions: Other: The calculation of blood IL-6 and coloctral milk melatonin
- women with elective cesarean section (Active Comparator): 30 women with elective cesarean section will be included in group 3serum IL-6 levels before and after delivery and colostral milk melatonin levels will be measured
  Interventions: Other: The calculation of blood IL-6 and coloctral milk melatonin

INTERVENTIONS:
Other: The calculation of blood IL-6 and coloctral milk melatonin — Collected maternal colostral milk will be sampled for melatonin levels.Blood samples driven before and after delivery will be evaluated for IL-6 levels in each group
  Other Names: No other intervention

SUMMARY:
The comparison of serum and colostral melatonin, and IL-6 levels between women with vaginal delivery, emergency cesarean section and elective cesarean section

DETAILED DESCRIPTION:
In this prospective randomized study, the investigators aimed to show the changes in the melatonin levels in colostral milk in spontaneous vaginal delivery,emergency cesarean and elective cesarean section patients and changes in blood IL-6 level before and after the delivery in same patient groups.

the investigators randomized 30 cases for each group for comparisons.Time range seems short in this study but participating hospital setting is a busy maternity hospital thus it will be performed easily.

The purpose of this study is to demonstrate the beneficial effect of spontaneous vaginal delivery on the secretion of melatonin which is solely secreted by the mother and the newborn is dependent on maternal milk oriented melatonin until 12 th week after delivery

ELIGIBILITY:
Inclusion Criteria

* Pregnant women reached term
* Patients with spontaneous vaginal delivery
* Patients preferred cesarean section electively
* Patient who had emergency cesarean section without additional medical or surgical problems

Exclusion Criteria

* Women who had history of intrauterine fetal loss
* Hypertention during pregnancy
* Anemia
* Thyroid diseases
* Patients with chronic diseases
* Smokers
* Drug users

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The serum IL-6 level | 8 weeks
  the measurement of serum IL-6 level in blood
Colostral Milk melatonin levels in different types of deliveries | 8 weeks
  Colostral milk taken from the postpartum midnight breast milk were evaluated for melatonin levels

CONTACTS AND LOCATIONS:
Overall Officials: Canan Soyer-Caliskan, Principal Investigator — Samsun EAH
Locations (1):
- Samsun EAH, Samsun, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No